CLINICAL TRIAL: NCT06618664
Title: A Randomized, Controlled, Open-label, Multicenter Phase III Clinical Study of Anti CTLA-4 Antibody SHR-8068 Combined With Adebrelimab and Bevacizumab Versus Sintilimab Combined With Bevacizumab for the First-line Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Study of SHR-8068 Combined With Adebrelimab and Bevacizumab Versus Sintilimab Combined With Bevacizumab for the Treatment of Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-8068-301
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — Bevacizumab; sintilimab

STUDY DESIGN:
Intervention Model Description: The study is a randomized, controlled, open-label phase III study designed for efficacy evaluation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-8068 combined with Adebrelimab and Bevacizumab (Experimental)
  Interventions: Drug: SHR-8068; Drug: Adebrelimab; Drug: Bevacizumab
- Sintilimab combined with Bevacizumab (Active Comparator)
  Interventions: Drug: Bevacizumab; Drug: Sintilimab

INTERVENTIONS:
Drug: SHR-8068 — SHR-8068: injection, 50 mg/10 mL, intravenous infusion
  Arms: SHR-8068 combined with Adebrelimab and Bevacizumab
Drug: Adebrelimab — Adebrelimab: injection, 600 mg/12 mL, intravenous infusion
  Arms: SHR-8068 combined with Adebrelimab and Bevacizumab
Drug: Bevacizumab — Bevacizumab: injection, 100 mg/4 mL, intravenous infusion
Drug: Sintilimab — Sintilimab: injection, 100 mg/10 mL, intravenous infusion
  Arms: Sintilimab combined with Bevacizumab

SUMMARY:
To evaluate the efficacy of SHR-8068 combined with Adebrelimab and Bevacizumab compared with Sintilimab combined with Bevacizumab for the first-line treatment of advanced HCC

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. ≥ 18 years old, both male and female
3. Unresectable locally advanced or metastatic HCC confirmed by histopathologically/cytologically
4. At least one measurable lesion based on RECIST v1.1 criteria
5. Barcelona clinic liver cancer: Stage B or C
6. No previous systemic antitumor therapy for HCC
7. ECOG PS of 0-1
8. Child-Pugh score of A or B7
9. Expected survival period ≥ 12 weeks
10. Adequate organ function
11. Blood pregnancy negative (women of childbearing age) and non-breastfeeding, effective contraception

Exclusion Criteria:

1. Hepatic cholangiocarcinoma, mixed hepatocellular carcinoma -cholangiocarcinoma, sarcomatoid hepatocellular carcinoma and fibrolamellar hepatocellular carcinoma
2. Patients with other malignancies currently or within the past 5 years
3. With known severe allergic reactions to any other monoclonal antibodies
4. Patients with known CNS metastasis or hepatic encephalopathy
5. Patients with liver tumor burden greater than 50% of total liver in volume or received liver transplants
6. Patients with symptomatic ascites or pleural effusion
7. Patients with hypertension which cannot be well controlled by antihypertensives
8. Uncontrolled cardiac diseases or symptoms
9. Known hereditary or acquired bleeding (e.g., coagulopathy) or a tendency to clot (e.g., hemophiliacs)
10. Major vascular disease occurred in the 6 months before randomization
11. Gastrointestinal perforation or gastrointestinal fistula within 6 months before randomization
12. Major surgery within 28 days before randomization or expected to require major surgery during the study period
13. Active infection, or fever of unknown cause ≥ 38.5℃ in the first 7 days of randomization, or WBC > 15×109/L at baseline
14. Known positive history of human immunodeficiency virus test or acquired immunodeficiency syndrome, known HBV infection, known HCV infection
15. Patients who received live vaccines within 28 days before randomization, or are expected to be vaccinated during the treatment period
16. Patients with other potential factors that may affect the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From Randomization to the first occurrence of disease progression as determined by the Blinded Independ Review Committee (BIRC) according to RECIST v1.1 or initiation of new anti-tumor therapy (up to approximately 36 months)
Overall survival (OS) | From randomization to death from any cause (whichever occurs first) (up to approximately 36 months)
  OS is defined as the time from randomization to death from any cause

SECONDARY OUTCOMES:
Time to Progression (TTP) | From randomization to the first occurrence of disease progression as determined by the Blinded Independ Review Committee (BIRC) according to RECIST v1.1 (up to approximately 36 months)]
  TTP is defined as the time from randomization to the until first evidence of disease progression as determined by the Blinded Independ Review Committee (BIRC) according to RECIST v1.1
Disease Control Rate (DCR) | From Randomization to the first occurrence of disease progression as determined by the Blinded Independ Review Committee (BIRC) according to RECIST v1.1 or initiation of new anti-tumor therapy (up to approximately 36 months)
  DCR is defined as the proportion of participants with Complete Response (CR), Partial Response (PR) or Stable Disease (SD), as determined by the Blinded Independ Review Committee (BIRC) according to RECIST v1.1
Objective Response Rate (ORR) | From Randomization to the first occurrence of disease progression or initiation of new anti-tumor therapy (up to approximately 36 months)
  ORR is defined as the proportion of participants with Complete Response (CR) or Partial Response (PR), as determined by the Blinded Independ Review Committee (BIRC) according to RECIST v1.1
Duration of Response (DoR) | From the first occurrence of a confirmed objective response to disease progression as determined by the Blinded Independ Review Committee (BIRC) according to RECIST v1.1 or death from any cause (whichever occurs first) (up to approximately 36 months)
  DOR is defined as the time from the first occurrence of a confirmed objective response to disease progression as determined by the Blinded Independ Review Committee (BIRC) according to RECIST v1.1 or death from any cause (whichever occurs first)
Time to Response (TTR) | From the first occurrence of complete response (CR) or partial response (PR) as determined by the Blinded Independ Review Committee (BIRC) according to RECIST v1.1 (up to approximately 36 months)
  TTR is defined as time from the randomization of Complete Response (CR) or Partial Response (PR) by the Blinded Independ Review Committee (BIRC) according to RECIST v1.1
The incidence, severity and relevance to investigational drugs of adverse events (AE) and serious adverse events (SAE) according to NCI-CTCAE v5.0 | From the ICF date until the end of the safety follow-up or initiation of new anti-tumor therapy (up to approximately 36 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided